CLINICAL TRIAL: NCT02433145
Title: Explore the Association Between Neuropsychological Functions and ADHD Diagnosis and Comorbid Using Longitudinal Study in Preschool Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201405086RINB
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD in preschoolers; neuropsychological functions; behavior inhibition; family function and parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The current study using the longitudinal study in preschool children to exam three study issues: 1) using the neuropsychological functions (ie. Behavioral inhibition, delay aversion, the variability of reaction time) among the preschool children predict the ADHD diagnosis and behavior symptoms in 1.5 years later. 2) using the behavior inhibition, delay aversion and the variability of reaction time (using the parameter among Gaussian distribution and ex-Gaussian distribution) explore the association between attention and motor inhibition problems. 3) explore the transaction effect between the neuropsychological functions and family function and parenting to predict ADHD comorbidity with oppositional defiant disorder.4) explore the association between the internalizing/ externalizing problems of ADHD and temperament. The current study has opportunity to describe and to answer the complicated problems for heterogeneous neuropsychological deficits in ADHD, and to elucidate the core issues for ADHD have comorbid with ODD. The most important contribution is to offer the empirical evidence to make a clean suggestion in ADHD diagnosis and intervention in preschool age.

DETAILED DESCRIPTION:
The current study would follow the same participants for 1.5 years, time 1 is around 4-5 years old, and time 2 is around 6-7 years old.

Participants:

* 100 typical developmental control
* 120 ADHD high risk preschool children at time 1

The diagnosis at time 2 to have three groups in this study:

* ADHD persistent
* ADHD remission
* typical developmental control

The measurements were included

* the different neuropsychological test (ie. behavioral inhibition, delay aversion, and vigilance task)
* the ADHD behavioral rating scales and diagnosis interview
* the scaling for family function and parenting
* intellectual assessment

This study could offer the suggestion for the further intervention in ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Control group

   * The subjects without ADHD.
   * Ages range from 4 to 5
   * Full scale IQ ≥ 80
   * The subjects who and whose parents consent to this study.
2. ADHD high risk group

   * Patients who have clinically diagnosis of DSM-IV ADHD confirmed by the Psychiatrists or have the risk of becoming ADHD confirmed by the ADHD behavioral rating scales.
   * Ages range from 4 to 5
   * Full scale IQ ≥ 80
   * Patients who and whose parents consent to this study.

Exclusion Criteria:

* Mental Retardation
* Schizophrenia, Schizoaffective Disorder
* Mood Disorders
* Organic Psychosis
* Learning Disorder
* Pervasive Developmental Disorder
* The subjects of control group if have a history of the following condition as defined by DSM-IV: ADHD in addition to the above exclusion criteria will be excluded.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will recruit 100 typical developmental control and 120 ADHD high risk preschool children at time 1, and we using the diagnosis at time 2 to have three groups in this study (ADHD persistent, ADHD remission and typical developmental control).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
The error rate and hit reaction time in the judgements on color flanker response inhibition test which measured by the e-prime program on the laptop | up to 3 years

SECONDARY OUTCOMES:
The error rate and hit reaction time in the day-night stroop test which measured by the e-prime program on the laptop | up to 3 years

OTHER OUTCOMES:
The final balloon numbers and eaction time in delay aversion test which measured by the e-prime program on the laptop | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan